CLINICAL TRIAL: NCT00785616
Title: A Trial to Determine the Long-term Durability of Virologic Suppression in Kaletra Recipients With Imperfect Adherence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Jonathan Shuter, Prof. Dept Medicine, Montefiore Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-03086E
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: HIV Infection
Keywords: HIV; Adherence; MEMS
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: MEMS cap monitoring — Electronic monitoring of medication adherence using MEMS caps
Other: MEMS cap monitoring — Adherence to antiretroviral medications will be measured using electronic bottle caps (MEMS caps) that record the time signature of each bottle opening.
Other: MEMS cap monitoring — Adherence to antiretroviral medications will be measured using electronic bottle caps (MEMS caps) that record the time/date signature of each bottle opening.

SUMMARY:
This study will enroll completers of a prior 24 week MEMS cap study of Kaletra adherence, conducted in 2005 - 2006, and repeat the MEMS monitoring for an additional 24 weeks in 2008/2009 on the current antiretroviral anchor drug. The goals of the study are to correlate long-term adherence with virologic outcome, and to explore the stability of MEMS cap adherence measurements over time.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the prior Kaletra MEMS cap study

Exclusion Criteria:

* Not receiving antiretroviral therapy, refusal to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Proportion with virologic suppression | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States